CLINICAL TRIAL: NCT06519708
Title: Analgesic Efficacy of Erector Spinae Plane Block vs External Oblique Intercostal Plane Block in Subcostal Cancer Surgeries: A Randomized Controlled Study
Brief Title: Analgesic Efficacy of Erector Spinae Plane Block vs External Oblique Intercostal Plane Block in Subcostal Cancer Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Osama Sayed Mohamed Ibrahim, Assistant Lecturer of Anesthesiology, Intensive Care Unit and Pain Medicine, Faculty of Medicine, Cairo University, Cairo, Egypt., National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AP2403-201-107
Record Dates: First submitted 2024-07-21; First posted 2024-07-25 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Analgesia; Erector Spinae Plane Block; External Oblique Intercostal Plane Block; Subcostal Cancer Surgeries
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane Block (Active Comparator): Patients will receive an ultrasound-guided erector spinae plane block with the injection of 30 ml bupivacaine 0.25% after induction of general anesthesia.
  Interventions: Drug: Erector Spinae Plane Block
- External Oblique Intercostal Plane Block (Experimental): Patients will receive an ultrasound-guided external oblique intercostal plan block Intraoperative with the injection of 30 ml bupivacaine 0.25% after induction of general anesthesia.
  Interventions: Drug: External Oblique Intercostal Plane Block

INTERVENTIONS:
Drug: Erector Spinae Plane Block — Patients will receive an ultrasound-guided erector spinae plane block with the injection of 30 ml bupivacaine 0.25% after induction of general anesthesia.
  Arms: Erector Spinae Plane Block
Drug: External Oblique Intercostal Plane Block — Patients will receive an ultrasound-guided external oblique intercostal plan block Intraoperative with the injection of 30 ml bupivacaine 0.25% after induction of general anesthesia.
  Arms: External Oblique Intercostal Plane Block

SUMMARY:
This study aims to evaluate the impact of ultrasound-guided erector spinae plane block compared to ultrasound-guided external oblique intercostal plane block regarding management of postoperative acute pain in patients undergoing above Umbilical surgical procedure.

DETAILED DESCRIPTION:
Subcostal incisions in cancer surgeries as in hepatectomy and nephrectomy are a cause of severe pain and can lead to significant respiratory impairment. Regional anesthesia of the trunk and abdominal wall is usually centered on epidural analgesia.

Erector spinae plane block (ESPB) is the deposition of local anesthetic (LA) in the interfascial plane at the paraspinal region. It provides effective visceral and somatic analgesia.

The recently described external oblique intercostal plane block (EOIPB) is a simple, effective, and convenient block, particularly in the context of morbid obesity, at which local anesthetic (LA) is deposited in the interfacial plane deep to external oblique muscle at the sixth intercostal space. It provides a blockade of the thoracoabdominal nerves at the level of T6 to T10.

ELIGIBILITY:
Inclusion Criteria:

* Age (18-65) Years.
* Both sexes.
* Body mass index (BMI): (20-40) kg/m2.
* American Society of Anesthesiology (ASA) physical status II, III.
* Type of surgery; unilateral subcostal incision in hepatectomy and nephrectomy.

Exclusion Criteria:

* Patient refusal.
* Subcostal incisions that are crossing the midline or midline incision.
* Age <18 years or >65 years
* BMI <20 kg/m2 and >40 kg/m2
* Known sensitivity or contraindication to drugs used in the study
* Contraindication to regional anesthesia e.g. local infection at the site of introduction, pre-existing peripheral neuropathies, and coagulopathy.
* Pregnancy.
* Physical status ASA IV
* patients on chronic analgesic therapy (daily morphine ≥30 mg or equivalent dose of other opioids or tramadol or any medication for neuropathic pain)
* patients with a history of drug abuse
* patients with neuropsychiatric diseases; patients with a history of chronic pain syndromes that may enhance sensitivity to pain, for example, fibromyalgia
* All patients who are going to have severe intra- or post-operative bleeding or will require postoperative mechanical ventilation are also excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-07-25 (Actual); Primary Completion 2026-01-10 (Actual); Study Completion 2026-01-17 (Actual)

PRIMARY OUTCOMES:
Total amount of morphine consumption | 24 hours postoperatively
  Rescue analgesia will be provided in the form of IV morphine 3 mg boluses if the patient indicates Numeric Pain Rating Scale ≥ 4. The total amount of morphine given in 24 hours will be recorded for the two groups. A maximum dose of 0.5 mg/kg/24hours of morphine is allowed.

SECONDARY OUTCOMES:
Total amount of intraoperative fentanyl consumption | Intraoperatively
  Rescue analgesia of fentanyl 1 μg/kg will be given if the mean arterial blood pressure or heart rate rises above 20% of baseline levels.
Heart rate | Till the end of surgery
  Heart rate will be recorded intraoperatively at 5-minute intervals till the end of surgery and the average of each three successive readings.
Mean arterial blood pressure | Till the end of surgery
  Mean arterial blood pressure will be recorded intraoperatively at 5-minute intervals till the end of surgery and the average of each three successive readings.
Time of first rescue analgesia | 24 hours postoperatively
  Time of first rescue analgesia will be recorded from the end of surgery to first dose of morphine administrated. Rescue analgesia will be provided in the form of IV morphine 3 mg boluses if the patient indicates Numeric Pain Rating Scale ≥ 4.
Complications | 24 hours postoperatively
  Complications related to blocks (local anesthetic systemic toxicity, pneumothorax and arterial puncture) and Morphine related complications (respiratory depression, urine retention or pruritis) will be recorded.
Patient satisfaction | 24 hours postoperatively
  Degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.